CLINICAL TRIAL: NCT00408746
Title: Prospective (Multicentre) Epidemiologic Longitudinal Study of Orofacial Development of Preterm and Low Birthweight Infants Compared to Term Infants in Consideration of Perinatal, Biometrical, Nutritional, Functional and Parental Parameters
Brief Title: Orofacial Development of Preterm and Low Birthweight Infants Versus Term Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: NUK Baby Care, Mapa GmbH, Industriestrasse 21-25, 27404 Zeven (Unknown); TOP-Service für Lingualtechnik GmbH, Lindenstr. 42, 49152 Bad Essen (Unknown)
Responsible Party: Priv.-Doz. Dr. Ariane Hohoff, University Hospital Muenster
Other Study IDs: KFO-MAPA-1/2006
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2007-02

CONDITIONS: Premature Birth; Infant, Newborn; Pregnancy
Keywords: stomatognathic system; maxilla; palate; development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: palatal development — Impressions of preterm and term palates.

SUMMARY:
Preterm infants account for 6 % of all live-births in western societies. Scientific evidence can be found for altered palatal morphology in the short term among preterm children. Oral intubation and orogastric feeding might be contributing factors to these alterations, but it has not been examined whether in the absence of these interventions preterm infants' palates are altered a priori as compared to term infants, e.g. due to immaturity of the bones or due to immaturity of oral function. Because of contradictory results, lack of longitudinal and high quality standard studies, the scientific evidence is also to weak to answer the question whether premature birth without or with a history of orotracheal intubation and orogastric feeding causes permanent alteration of orofacial development. The aim of the present study, therefore is to investigate in consideration of perinatal, biometrical, nutritional, functional and parental parameters.

DETAILED DESCRIPTION:
Preterm infants account for 6 % of all live-births in western societies. Scientific evidence can be found for altered palatal morphology in the short term among preterm children. Oral intubation and orogastric feeding might be contributing factors to these alterations, but it has not been examined whether in the absence of these interventions preterm infants' palates are altered a priori as compared to term infants, e.g. due to immaturity of the bones or due to immaturity of oral function. Because of contradictory results, lack of longitudinal and high quality standard studies, the scientific evidence is also to weak to answer the question whether premature birth without or with a history of orotracheal intubation and orogastric feeding causes permanent alteration of orofacial development.

The aim of the present study, therefore is to investigate in consideration of perinatal, biometrical, nutritional, functional and parental parameters

* whether preterm babies without a history of orotracheal intubation and orogastric feeding do have an altered orofacial development as compared to term babies.
* in a second step whether preterm babies with a history of orotracheal intubation and orogastric feeding do have an altered orofacial development as compared to preterm and term infants without these interventions.

The participants must meet the following inclusion criteria:

all:

* caucasian origin and
* informed consent by both parents. term infants:
* born at ≥ 37 weeks of gestation
* birthweight ≥ 2500 g.

preterm infants (will be allocated in two groups depending on the absence or presence of a history of orotracheal intubation and orogastric feeding):

* gestational age at birth > 25 weeks and
* birthweight > 500 g.

Exclusion criteria are hydrocephalus, oral or facial clefts, congenital syndrome, deformity of the head and neck and congenital metabolic disease beyond osteopenia of prematurity.

The children will be examined at the following times:

* 2-5 days prior to discharge from hospital (weight > 1800 g in the preterm group)
* 40 weeks of gestation ( + 7 days tolerance)
* 3, 6, 9, 12, 15 and 18 months of corrected age (+ 28 days tolerance)
* 24, 36, 48 and 60 months of corrected age (+ 28 days tolerance).

The following measures will be taken at all times:

child:

* standardized questionnaire for evaluation of biometrical (weight, length/height, head circumference), nutritional and functional parameters (breast/bottle/spoon feeding, mode of breathing, lip and tongue posture, sucking habits, kind of pacifiers and suckers)
* standardized frontal and lateral photographs
* alginate impressions of the upper jaw
* measurement of the overjet.

child and parents: - smear of the oral mucosa.

The following measures will be taken once (at time of discharge from hospital):

child:

* standardized questionnaire concerning perinatal parameters. parents:
* standardized questionnaire concerning parents orofacial history
* standardized frontal and lateral photographs
* alginate impressions of the both jaws and wax bite
* measurement of the overjet
* dental and periodontal findings.

The following measures will be taken at the investigation times during the time the child is breast or bottle fed (measures stopped at the latest when the child has a corrected age of twelve months:

child:

* sucking of the child at an alginate filled condom
* ultrasound of the feeding process.

The following measures will be taken at a corrected age of 36 and 50 months:

child:

- alginate impression of the lower jaw, wax bite.

As a positive side effect the database -beyond the primary aim of the study- will be useful in evaluating the influence of hereditary, perinatal, functional and nutritional parameters on orofacial development in general, it will serve as control data for therapies in patients with craniofacial defects (e.g. clefts) and provide a basis for development of physiologic pacifying, feeding and intensive care devices.

ELIGIBILITY:
Inclusion Criteria:

* infants of the tertiary care level University Hospital of Münster
* delivery between May 1999 and December 2008
* caucasian origin
* written informed consent by both parents

Exclusion Criteria:

* history of orotracheal intubation / orogastric tube feeding
* hydrocephalus
* palatal cleft, congenital syndrome, head / neck malformation
* congenital metabolic disease beyond osteopenia of prematurity

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Caucasian preterm and term babies
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2003-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Hohoff, PD Dr., Principal Investigator — Universitätsklinikum Münster, Germany
Locations (1):
- Universitätsklinikum Münster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Hohoff A, Rabe H, Ehmer U, Harms E. Palatal development of preterm and low birthweight infants compared to term infants - What do we know? Part 1: The palate of the term newborn. Head Face Med. 2005 Oct 28;1:8. doi: 10.1186/1746-160X-1-8. PMID 16270908
- [Background] Hohoff A, Rabe H, Ehmer U, Harms E. Palatal development of preterm and low birthweight infants compared to term infants - What do we know? Part 2: The palate of the preterm/low birthweight infant. Head Face Med. 2005 Oct 28;1:9. doi: 10.1186/1746-160X-1-9. PMID 16270909
- [Background] Hohoff A, Rabe H, Ehmer U, Harms E. Palatal development of preterm and low birthweight infants compared to term infants -- What do we know? Part 3: discussion and conclusion. Head Face Med. 2005 Nov 2;1:10. doi: 10.1186/1746-160X-1-10. PMID 16270912
- [Background] Hohoff A, Stamm T, Meyer U, Wiechmann D, Ehmer U. Objective growth monitoring of the maxilla in full term infants. Arch Oral Biol. 2006 Mar;51(3):222-35. doi: 10.1016/j.archoralbio.2005.07.007. Epub 2005 Aug 31. PMID 16139239